CLINICAL TRIAL: NCT05319899
Title: A Phase 1, Single-Center, Randomized, 3-Period Crossover Study to Evaluate the Relative Bioavailability of WTX101 in Healthy Subjects After Single Dose Administration of a Non-Coated Formulation With and Without a Proton Pump Inhibitor and With a Proton Pump Inhibitor With and Without Food
Brief Title: A Study of ALXN1840 (Non-coated) Administered With And Without Omeprazole In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: WTX101-101; CA12887 (Other: Celerion)
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: ALXN1840; WTX101; Omeprazole
MeSH Terms: interventions — rhoA GTP-Binding Protein; tetrathiomolybdate; Omeprazole

STUDY DESIGN:
Intervention Model Description: This was single-center, open-label, randomized, 3-period, 3-treatment, 6-sequence crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1: ABC (Experimental): Participants received each treatment on 1 occasion:
  Period 1 (Treatment A): ALXN1840 following an overnight fast. Period 2 (Treatment B): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, following an overnight fast. Period 3 (Treatment C): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840; Drug: Omeprazole
- Sequence 2: ACB (Experimental): Participants received each treatment on 1 occasion:
  Period 1 (Treatment A): ALXN1840 following an overnight fast. Period 2 (Treatment C): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 3 (Treatment B): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840; Drug: Omeprazole
- Sequence 3: BAC (Experimental): Participants received each treatment on 1 occasion:
  Period 1 (Treatment B): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, following an overnight fast. Period 2 (Treatment A): ALXN1840 following an overnight fast. Period 3 (Treatment C): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840; Drug: Omeprazole
- Sequence 4: BCA (Experimental): Participants received each treatment on 1 occasion:
  Period 1 (Treatment B): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, following an overnight fast. Period 2 (Treatment C): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 3 (Treatment A): ALXN1840 following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840; Drug: Omeprazole
- Sequence 5: CAB (Experimental): Participants received each treatment on 1 occasion:
  Period 1 (Treatment C): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 2 (Treatment A): ALXN1840 following an overnight fast. Period 3 (Treatment B): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840; Drug: Omeprazole
- Sequence 6: CBA (Experimental): Participants received each treatment on 1 occasion:
  Period 1 (Treatment C): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 2 (Treatment B): Omeprazole once daily in the morning of Days -5 to -1 following an overnight fast, omeprazole at Hour -1 on Day 1 following an overnight fast, and ALXN1840 at Hour 0 on Day 1, following an overnight fast. Period 3 (Treatment A): ALXN1840 following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840; Drug: Omeprazole

INTERVENTIONS:
Drug: ALXN1840 — ALXN1840 (60 milligrams) was administered orally as non-coated capsules at Hour 0 on Day 1.
  Other Names: WTX101 (formerly); Bis-choline tetrathiomolybdate; Tiomolibdate choline
Drug: Omeprazole — Omeprazole (20 milligrams) was administered orally as a delayed-release capsule in the morning of Days -5 to -1 and at Hour -1 on Day 1.
  Other Names: Prilosec

SUMMARY:
This was single-center, open-label, randomized, 3-period, 3-treatment, 6-sequence crossover study evaluating the PK of single doses of WTX101 in healthy participants based on the measurement of plasma total Molybdenum.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* Medically healthy with no clinically significant laboratory profiles, vital signs, or electrocardiograms.
* Body mass index ≥ 18 and ≤ 32.0 kilograms/meter squared.
* Willing and able to adhere to contraception requirements.

Exclusion Criteria:

* Participant was mentally or legally incapacitated
* History or presence of clinically significant medical or psychiatric condition or disease.
* History of any illness that might have interfered with drug absorption.
* History or presence of hypersensitivity or idiosyncratic reaction to the study medications, study medication excipients.
* History or presence of alcoholism or drug abuse.
* Female participants who were pregnant or lactating.
* Positive results at screening for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus.
* Serum ceruloplasmin and copper values outside of the normal range at screening.
* On a diet incompatible with the on-study diet within the 28 days prior to the first ALXN1840 dose and throughout the study; unable to consume the contents of a high-fat breakfast.
* Participation in a previous clinical trial with ALXN1840.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2014-03-24 (Actual); Study Completion 2014-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to one of 6 treatment sequences.
Groups:
- Treatment Sequence 1: ABC: Participants received each treatment on 1 occasion:
  Period 1 (Treatment A): ALXN1840 60 milligrams (mg) (2 x 30 mg capsules) on Day 1 following an overnight fast. Period 2 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) once daily (QD) in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast. Period 3 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
- Treatment Sequence 2: ACB: Participants received each treatment on 1 occasion:
  Period 1 (Treatment A): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast. Period 2 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 3 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
- Treatment Sequence 3: BAC: Participants received each treatment on 1 occasion:
  Period 1 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast. Period 2 (Treatment A): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast. Period 3 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
- Treatment Sequence 4: BCA: Participants received each treatment on 1 occasion:
  Period 1 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast.
  Period 2 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 3 (Treatment A): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
- Treatment Sequence 5: CAB: Participants received each treatment on 1 occasion:
  Period 1 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 2 (Treatment A): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast. Period 3 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
- Treatment Sequence 6: CBA: Participants received each treatment on 1 occasion:
  Period 1 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast. Period 2 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast. Period 3 (Treatment A): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
Period: Overall Study
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: ACB | Treatment Sequence 3: BAC | Treatment Sequence 4: BCA | Treatment Sequence 5: CAB | Treatment Sequence 6: CBA
Started | 3 | 3 | 3 | 3 | 3 | 3
Received at Least 1 Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Treatment Sequence 1: ABC: Participants received each treatment on 1 occasion:
  Period 1 (Treatment A): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast. Period 2 (Treatment B): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast. Period 3 (Treatment C): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: ACB | Treatment Sequence 3: BAC | Treatment Sequence 4: BCA | Treatment Sequence 5: CAB | Treatment Sequence 6: CBA | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (4.16) | 31.3 (10.21) | 25.7 (2.52) | 36.0 (14.11) | 35.0 (17.69) | 40.0 (12.53) | 33.1 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 2 | 2 | 1 | 9
  Male | 3 | 2 | 0 | 1 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of Total Molybdenum (Mo)
Description: AUC0-t was calculated by the linear trapezoidal method.
Time Frame: Predose (0 hour) up to 192 hours postdose
Population: Pharmacokinetic (PK) analysis population included all participants who completed at least 2 periods of the study and had sufficient data for the determination of PK parameters.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Groups:
- Treatment A: ALXN1840 (Fasted): ALXN1840 60 mg (2 x 30 mg capsules) on Day 1 following an overnight fast.
- Treatment B: Omeprazole + ALXN1840 (Fasted): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, following an overnight fast.
- Treatment C: Omeprazole + ALXN1840 (Fed): Omeprazole 20 mg (1 x 20 mg delayed-release capsule) QD in the morning of Days -5 to -1 following an overnight fast, omeprazole 20 mg at Hour -1 on Day 1 following an overnight fast, and ALXN1840 60 mg (2 x 30 mg capsules) at Hour 0 on Day 1, approximately 30 minutes after the start of a high-fat breakfast.
Arm/Group | Treatment A: ALXN1840 (Fasted) | Treatment B: Omeprazole + ALXN1840 (Fasted) | Treatment C: Omeprazole + ALXN1840 (Fed)
Number analyzed (Participants) | 18 | 18 | 18
hours*ng/mL | 14531 (6886) | 18537 (4303) | 14536 (3663)
Statistical Analysis 1: Comparison: Treatment A: ALXN1840 (Fasted) vs Treatment B: Omeprazole + ALXN1840 (Fasted); Analysis was performed using analysis of variance (ANOVA); Test type: Other; Geometric Mean Ratio (%) = 140.63, 90% CI 2-sided [118.94 to 166.26]
Statistical Analysis 2: Comparison: Treatment B: Omeprazole + ALXN1840 (Fasted) vs Treatment C: Omeprazole + ALXN1840 (Fed); Analysis was performed using ANOVA; Test type: Other; Geometric Mean Ratio (%) = 77.65, 90% CI 2-sided [65.67 to 91.80]

2. Primary Outcome: Maximum Measured Plasma Concentration (Cmax) of Total Mo
Time Frame: Predose (0 hour) up to 192 hours postdose
Population: PK analysis population included all participants who completed at least 2 periods of the study and had sufficient data for the determination of PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A: ALXN1840 (Fasted) | Treatment B: Omeprazole + ALXN1840 (Fasted) | Treatment C: Omeprazole + ALXN1840 (Fed)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 330 (124) | 401 (78.3) | 385 (71.3)
Statistical Analysis 1: Comparison: Treatment A: ALXN1840 (Fasted) vs Treatment B: Omeprazole + ALXN1840 (Fasted); Analysis was performed using ANOVA; Test type: Other; Geometric Mean Ratio (%) = 128.23, 90% CI 2-sided [112.99 to 145.52]
Statistical Analysis 2: Comparison: Treatment B: Omeprazole + ALXN1840 (Fasted) vs Treatment C: Omeprazole + ALXN1840 (Fed); Analysis was performed using ANOVA; Test type: Other; Geometric Mean Ratio (%) = 95.94, 90% CI 2-sided [84.54 to 108.88]

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered with the study drug and which did not necessarily have a causal relationship with the study drug. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A TEAE was defined as an AE that started or worsened at the time of or after study drug administration. An AE that occurred during the washout period between drugs was considered treatment emergent to the last drug given. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 through 14 days following final dose (up to Day 43)
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: ALXN1840 (Fasted) | Treatment B: Omeprazole + ALXN1840 (Fasted) | Treatment C: Omeprazole + ALXN1840 (Fed)
Number analyzed (Participants) | 18 | 18 | 18
Participants | 6 | 5 | 6

ADVERSE EVENTS:
Time Frame: Day 1 through 14 days following final dose (up to Day 43)
Description: All enrolled participants who received at least 1 dose of study drug.
Arm/Group | Treatment A: ALXN1840 (Fasted) | Treatment B: Omeprazole + ALXN1840 (Fasted) | Treatment C: Omeprazole + ALXN1840 (Fed)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 6/18 | 5/18 | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: ALXN1840 (Fasted) (N=18) | Treatment B: Omeprazole + ALXN1840 (Fasted) (N=18) | Treatment C: Omeprazole + ALXN1840 (Fed) (N=18)
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes